CLINICAL TRIAL: NCT02463331
Title: Possible Role of Chloroquine in Conjunction to Prednisone to Induce a Complete Remission in the Treatment of Autoimmune Hepatitis: a Randomized Trial
Brief Title: Possible Role of Chloroquine to Induce a Complete Remission in the Treatment of Autoimmune Hepatitis: a Randomized Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Lydia Teófilo de Moraes Falcão, Association of Chloroquine and Prednisone as an Alternative Treatment for Autoimmune Hepatitis: a Randomized Trial, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0571/04
Record Dates: First submitted 2015-05-18; First posted 2015-06-04 (Estimated); Results first posted 2016-12-30 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: Autoimmune Hepatitis
Keywords: autoimmune hepatitis; chloroquine; treatment
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — chloroquine diphosphate; Chloroquine; Prednisone; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chloroquine plus prednisone (Active Comparator): Chloroquine diphosphate 250mg/day associated to prednisone in variable doses
  Interventions: Drug: Chloroquine diphosphate; Drug: prednisone
- azathioprine plus prednisone (Experimental): azathioprine in variable doses (50-150mg/day) associated to prednisone in variable doses
  Interventions: Drug: prednisone; Drug: azathioprine

INTERVENTIONS:
Drug: Chloroquine diphosphate — One pill of chloroquine diphosphate per day until the end of the study
  Other Names: Chloroquine
  Arms: chloroquine plus prednisone
Drug: prednisone — Prednisone 5-15 mg/day until the end of the study
Drug: azathioprine — azathioprine 1-2mg/Kg/day until the end of the study
  Arms: azathioprine plus prednisone

SUMMARY:
The gold-standard treatment of Autoimmune hepatitis (AIH), with prednisone alone or in conjunction with azathioprine can reach resolution of the disease in 70-80% of the cases in US. However, in Brazil the response to these treatments seems to be worse, approximately 35% in five years. Because of the side effects of the gold-standard treatment and the need for an alternative option for the no responsive patients, news drugs must be evaluated for this proposal. Chloroquine diphosphate is an antimalarial drug that has been used for the treatment of rheumatological diseases for at the least five decades. Chloroquine was used as a single drug for up to two years for the maintenance of AIH remission in an open study. There was a 6.49 greater chance of relapse in the historical controls when compared with patients treated with chloroquine (72.2% x 23.5%; p = 0.031). The aim of this study was to investigate whether chloroquine in conjunction with prednisone can be used as an alternative treatment of AIH in a randomized study, and to evaluate its side effects.

DETAILED DESCRIPTION:
Autoimmune hepatitis (AIH) is a chronic disease with a progressive destruction of hepatic parenchyma, leading to cirrhosis and high mortality in the absence of specific treatment. It has been demonstrated that the treatment with corticosteroids and azathioprine provides clinical and laboratory improvement, reduction of histological inflammatory activity on liver biopsy and an increased survival.

Because of the side effects of the gold-standard treatment and the need for an alternative option for the no responsive patients, news drugs must be evaluated for this proposal.

Chloroquine is a drug of the group of 4-aminoquinolines, synthetic derivatives of quinine and constituent of the bark of the Cinchona tree. Chloroquine accumulates in tissues in considerable amounts. In animals, from 200 to 700 times the plasma concentration can be found in liver, spleen, kidneys and lungs. As a weak base, it accumulates intracellularly, particularly in lysosomes with a consequent increase in pH within these organelles, which could contribute to its toxicity. Lysosomal lamellar bodies are observed in tissues affected by chloroquine, such as retina and neuromuscular system. Chloroquine inhibits the absorption and the binding of mitochondrial calcium, alters the membrane permeability and the transport of enzymes to the lysosomes. Apparently there are other mechanisms to explain its anti-inflammatory action; such as the interference with the release of TNF from mononuclear phagocytes by inhibiting gene expression and the down-regulation of TNF receptors, by delaying their transport to the cellular surface. Due to these mechanisms of action, chloroquine has anti-inflammatory activities and therefore is used in diseases such as rheumatoid arthritis and systemic lupus erythematosus. In liver diseases, chloroquine was used in patients with hepatitis B with normalization of the levels of aminotransferases and of the prothrombin time during treatment and relapse after drug discontinuation. Chloroquine was also evaluated in patients with porphyria cutanea tarda and despite the clinical and biochemical improvement, liver biopsies remained unchanged after one year of treatment.

A previous pilot study was performed in our institution, and published in 2005, with chloroquine diphosphate for the maintenance treatment of AIH. In this study, 14 patients with a biochemical and histological remission were treated with chloroquine diphosphate 250 mg/day for at least 12 months or until disease recurrence, and compared with 18 historical controls, which was held in discontinuation of treatment after remission. The chance of relapse was 6.49 times higher in the historical controls when compared with patients in the group treated with chloroquine (72.2% versus 23.5%, p = 0.031). The use of chloroquine was safe in patients with liver cirrhosis without decompensation, and there were no serious adverse events within two years of use.

The most common adverse effects of chloroquine are mild and transient such as gastrointestinal symptoms, headache, dizziness, blurry vision and fatigue. The more severe reactions described are itching, cardiovascular manifestations, dyskinesias, eye injuries, neuromuscular disorders and hearing loss. Among the most feared adverse effects of chloroquine, are the eye injuries, usually associated with chronic treatment. They may consist of changes in the retina, lens, cornea and optic nerve. Usually they remain stable after drug withdrawal, if the drug is discontinued in early stages. However, the retinal damage can increase when found in advanced stages, and may progress even years after cessation of chloroquine. It is believed that the chloroquine retinopathy can be prevented or recognized in an early reversible stage with judicious use, appropriate doses and regular ophthalmologic follow-up. It is recommended that the daily dose does not exceed 250 mg of chloroquine diphosphate or 400 mg of hydroxychloroquine, and ophthalmologic evaluations are carried out every 4 to 6 months. Despite the adverse effects and toxic reactions described above, there is a consensus in most studies with chloroquine that it is a well tolerated drug, provided that the appropriate dosage guidelines and regular eye examinations are followed. With these cautions in mind, its use rarely causes serious side or irreversible effects.

The aim of this study was to investigate whether chloroquine in conjunction with prednisone can be used as an alternative treatment of AIH in a randomized study, and to evaluate its side effects.

To be included patients had to satisfy the following criteria simultaneously: a diagnosis of probable / definite AIH and the indication of treatment (according to the International AIH Group), normal liver function and absence of clinical signs of decompensated liver disease (ascites, hepatic encephalopathy, gastrointestinal bleeding and hepatocellular carcinoma). For their enrollment, it is necessary that the patients are in accordance with the proposed study, following the precepts of the Declaration of Helsinki. If patients refuse to participate in the study, they will be treated following the traditional guidelines of our service. Treatment will be discontinued in case of pregnancy, patient's desire, side-effects or relapse of AIH.

Patients were randomized to receive azathioprine and prednisone or chloroquine and prednisone. The alternative treatment, with chloroquine, was maintained unless it caused major side-effects, no biochemical response or treatment failure. In this case, azathioprine was introduced in association with prednisone. All patients had visits every 30 days during the first six months with routine blood tests performed. After then, consultations were every two months. All complaints were recorded. Every patient were treated by the doctors responsible for the study, laboratory tests were performed in the Central Laboratory of the hospital. All patients underwent to initial ophthalmologic evaluation followed by six-monthly evaluations. The drug was withdrawal, if changes suggestive of retinopathy were observed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autoimmune hepatitis according to Autoimmune Hepatitis International Group with indication for treatment
* No evidence of decompensated liver cirrhosis
* Non-pregnant women and women with no intention to become pregnant
* Willing to participate in the study

Exclusion Criteria:

* Discrete biochemical changes and histological inflammatory activity absent / minimal (periportal / peri-septal: 0/1 +) or decompensated cirrhosis
* Cases of loss of follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2003-05; Primary Completion 2015-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo LR Cançado, Principal Investigator — University of Sao Paulo General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] T de Moraes Falcao L, Terrabuio DRB, Diniz MA, da Silva Evangelista A, Souza FG, R Cancado EL. Efficacy and safety of chloroquine plus prednisone for the treatment of autoimmune hepatitis in a randomized trial. JGH Open. 2019 Sep 10;4(3):371-377. doi: 10.1002/jgh3.12258. eCollection 2020 Jun. PMID 32514439

RESULTS

PARTICIPANT FLOW:
Groups:
- Azathioprine Plus Prednisone: azathioprine in variable doses (1-2mg/Kg/day) associated to prednisone in variable doses
  prednisone: Prednisone 5-15 mg/day until the end of the study
  azathioprine: azathioprine 1-2mg/Kg/day until the end of the study
Period: Overall Study
Arm/Group | Chloroquine Plus Prednisone | Azathioprine Plus Prednisone
Started | 26 | 31
Completed | 10 | 25
Not Completed | 16 | 6
Not completed — Adverse Event | 4 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Pregnancy | 2 | 3
Not completed — Lack of Efficacy | 6 | 0
Not completed — Physician Decision | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chloroquine Plus Prednisone | Azathioprine Plus Prednisone | Total
Number analyzed (Participants) | 26 | 31 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.54 (15.99) | 37.23 (17.63) | 37.28 (16.84)
Gender [Count of Participants; unit: Participants]
  Female | 21 | 24 | 45
  Male | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Response to Therapy
Description: The biochemical response is defined when there is normalization of hepatic enzymes, mainly AST and ALT.
Time Frame: six months
Measure: Count of Participants; unit: Participants
Arm/Group | Chloroquine Plus Prednisone | Azathioprine Plus Prednisone
Number analyzed (Participants) | 26 | 31
Participants | 14 | 21

2. Secondary Outcome: Histopathological Response to Therapy
Description: Histopathological response is achieved when there is minimal or no inflammation in hepatic tissue, as assessed by liver biopsy.
Time Frame: liver biopsy was was performed to evaluate histopathological response after 18 months of biochemical response
Population: The histological response was only evaluated in the patients with biochemical remission, since in the patients without biochemical response it was already known that there would be activity in the liver tissue.
Measure: Count of Participants; unit: Participants
Arm/Group | Chloroquine Plus Prednisone | Azathioprine Plus Prednisone
Number analyzed (Participants) | 14 | 21
Participants | 4 | 10

ADVERSE EVENTS:
Arm/Group | Chloroquine Plus Prednisone | Azathioprine Plus Prednisone
Serious Adverse Events (participants affected / at risk) | 6/26 | 0/31
Other Adverse Events (participants affected / at risk) | 3/26 | 2/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chloroquine Plus Prednisone (N=26) | Azathioprine Plus Prednisone (N=31)
machulopatia (Eye disorders) | 6 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chloroquine Plus Prednisone (N=26) | Azathioprine Plus Prednisone (N=31)
hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 1
gastric intolerance (Gastrointestinal disorders) | 0 | 1
neuropathy (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No